CLINICAL TRIAL: NCT04574973
Title: Optimizing Transcranial Direct Current Stimulation for Motor Recovery From Severe Post-stroke Hemiparesis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Relocation of PI
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 47644
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Hemiparesis
Keywords: neuroplasticity; rehabilitation; transcranial direct current stimulation; motor training
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anodal tDCS (Experimental): Subjects will receive 20 minutes of active, excitatory transcranial direct current stimulation of the ipsilesional hemisphere at 1.4mA, followed by 2 hours of intensive motor therapy of the affected upper extremity.
  Interventions: Device: transcranial direct current stimulation; Behavioral: intensive upper extremity motor training
- Cathodal tDCS (Experimental): Subjects will receive 20 minutes of active, excitatoryinhibitory transcranial direct current stimulation of the contralesional hemisphere at 1.4mA, followed by 2 hours of intensive motor therapy of the affected upper extremity.
  Interventions: Device: transcranial direct current stimulation; Behavioral: intensive upper extremity motor training
- Dual tDCS (Experimental): Subjects will receive 20 minutes of active, excitatory transcranial direct current stimulation of the ipsilesional hemisphere and inhibitory transcranial direct current stimulation of the contralesional hemisphere at 1.4mA, followed by 2 hours of intensive motor therapy of the affected upper extremity.
  Interventions: Device: transcranial direct current stimulation; Behavioral: intensive upper extremity motor training
- Sham tDCS (Sham Comparator): Subjects will receive 20 minutes of sham transcranial direct current stimulation, followed by 2 hours of intensive motor therapy of the affected upper extremity.
  Interventions: Device: transcranial direct current stimulation; Behavioral: intensive upper extremity motor training

INTERVENTIONS:
Device: transcranial direct current stimulation — This is a non-invasive form of stimulation which delivers safe, low levels of electrical current to the brain through the scalp.
Behavioral: intensive upper extremity motor training — This training is administered one-on-one with an occupational therapist. Activities will be focused on skills to help the individual function better in daily life.

SUMMARY:
Individuals who experienced a stroke over one year ago will be randomly assigned to receive 1 of 4 different conditions of brain stimulation. All individuals will receive therapy of the hand and arm following the stimulation. This study will try to determine which brain stimulation condition leads to the greatest improvement in hand and arm function.

DETAILED DESCRIPTION:
This study will look at the effects of a painless, non-invasive form of brain stimulation, called transcranial direct current stimulation, or tDCS. tDCS is thought to increase the brain's ability to change. Participants will be assigned to one of four groups by chance. Three groups will receive tDCS at a level expected to increase the brain's ability to change, and will vary by the areas of the brain that are stimulated. The fourth group will receive tDCS at a level not thought to affect the brain's ability to change. All participants will receive intensive therapy of their impaired arm and hand, focusing on exercises that will improve their ability to function in daily life.

ELIGIBILITY:
Inclusion Criteria:

* 12 or more months post-stroke
* Inability to extend the affected metacarpophalangeal joints at least 10 degrees and the wrist 20 degrees

Exclusion Criteria:

* Addition or change in dosage of drugs known to exert detrimental effects on motor recovery within 3 month of enrollment
* Untreated depression
* History of multiple strokes

Exclusion criteria for TMS evaluations:

* History of head injury with loss of consciousness
* History of severe alcohol or drug abuse, or psychiatric illness
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Presence of ferromagnetic material in the cranium except in the mouth, including metal fragments from occupational exposure and surgical clips in or near the brain
* Cardiac or neural pacemakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2021-01-08 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment from baseline | Baseline, Immediately post-intervention, one-month follow-up
  This provides a quantitative measure of motor recovery, balance, sensation, coordination, and speed. An increase in score indicates an improvement in function.

SECONDARY OUTCOMES:
Change in Action Research Arm Test from baseline | Baseline, Immediately post-intervention, one-month follow-up
  This consists of 4 tests to measure grasp, grip, pinch, and gross movement. An increase in score indicates an improvement in function.
Change in Stroke Impact Scale from baseline | Baseline, Immediately post-intervention, one-month follow-up
  This is a self-report measure of 64 items that assess 8 domains, including strength, hand function, activities of daily living, mobility, communication, emotion, memory and thinking, and participation. A score increase indicates an improvement.
Change in cortical motor map from baseline | Baseline, Immediately post-intervention, one-month follow-up
  This is performed using non-invasive transcranial magnetic stimulation to determine which parts of the brain control a muscle in the arm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky at Cardinal Hill Rehabilitation Hospital, Lexington, Kentucky, United States